CLINICAL TRIAL: NCT00305123
Title: The Molecular Epidemiology of Streptococcus Pyogenes Among Children in Bamako, Mali (Bamako BGAS2000)
Brief Title: Molecular Epidemiology of Streptococcus Pyogenes Among Children in Bamako, Mali
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 06-0002; Bamako BGAS2000
Record Dates: First submitted 2006-03-17; First posted 2006-03-21 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2009-10

CONDITIONS: Streptococcus Group A
Keywords: Pharyngitis, Mali, Group A Streptococcus, Children
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — GAS isolates.

GROUPS / COHORTS (1):
- 1: 12,000 children 5 to 16 years of age attending the 4 public elementary schools in Djikoroni-para-Sébénikoro, Bamako, Mali.

SUMMARY:
The purpose of this study is to learn more about sore throats caused by the germ Group A Streptococcus (GAS) or "Strep". When "Strep" causes a sore throat, it can be treated with medicines called antibiotics. However, if not treated, it can lead to heart problems and other serious diseases. This study will identify the different types of "Strep" that are present in children with sore throats. Researchers will check children with sore throats at least twice weekly among a group of approximately 12,000 children. Study participants will include children, ages 5-16, attending the public elementary schools in Djikoroni-Sébénikoro, a low income community in Bamako, Mali. Throat swabs will be obtained and free treatment is available when a child enrolled in the group complains of a sore throat. The information from this study may help make a vaccine to prevent "Strep" infection in Malian children. Children may participate for the 3 year duration of the study.

DETAILED DESCRIPTION:
Data on the epidemiology of group A streptococci (GAS) infection in developing countries is limited. Available publications suggest that not only is disease prevalent, but severe manifestations continue to occur at a high rate. Several promising GAS vaccine candidates are in pre-clinical and clinical development. One approach that has entered clinical trial is the use of a multivalent recombinant fusion peptide vaccine containing amino-terminal M protein fragments. In animal models, these M-protein type-specific epitopes induce protective opsonic antibodies that do not cross-react with human tissues. If type-specific vaccines are to be used in developing countries, then the molecular epidemiology of GAS in these settings must be better characterized. The primary objective of this study is to identify the genotypes (emm type or sub-type) of GAS isolated from 5 to 16 year old schoolchildren with pharyngitis living in a poor urban community in Bamako, Mali. The secondary objectives are: to characterize the molecular epidemiology of GAS pharyngitis among Malian schoolchildren by determining the distribution of genotypes according to age in years, year of study, and season (cold or dry); to estimate the incidence of GAS pharyngitis among 5 to 16 year old schoolchildren living in a poor urban community in Bamako, Mali overall and by age, gender, year of study, and season; and to describe the clinical features of GAS pharyngitis among the Malian schoolchildren. Surveillance for pharyngitis will be conducted at least twice weekly among a cohort of approximately 12,000 children, ages 5-16, attending the four public elementary schools in Djikoroni-para-Sébénikoro, a low-income community in Bamako, Mali. Throat swabs will be obtained when a child enrolled in the cohort complains of a sore throat. GAS isolated from the swabs will be characterized by emm typing. The primary endpoint of the study is the proportion of each emm-type among children with GAS pharyngitis. The secondary endpoints include the following: the proportion of each emm-type among children with GAS pharyngitis overall and according to age in years, year of study, and season (cold or dry); the proportion of children with pharyngitis from whom GAS is isolated; the minimal incidence of GAS pharyngitis per 100,000 children in the catchment area of Djikoroni-para-Sébénikoro overall and according to: age in years, gender, year of study, and season (cold or dry); the incidence density (number of cases per children-weeks of follow up) of GAS pharyngitis among enrolled school children overall and according to: age in years, year of study, and season (cold or dry); and the proportion of children with GAS pharyngitis who experience symptoms such as fever, exudative pharyngitis, tender cervical adenopathy, or scarletiniform rash, overall and by age in years. It is clear that GAS is an important worldwide pathogen and that it has been understudied in much of the developing world. Given the early successes of multivalent M type-specific vaccines, investigations of the molecular epidemiology delineating the distribution of the emm-types of the organism associated with pharyngitis (and therefore presumably acute rheumatic fever) are crucial for designing a vaccine that has utility in preventing rheumatic heart disease and other GAS disease in the developing world. The current protocol is intended to provide data to address these goals.

ELIGIBILITY:
Inclusion Criteria:

* 5 to 16 years old (at enrollment/beginning of the school year).
* Enrolled at one of the 4 participating elementary schools in Djikoroni-para/Sébénikoro.
* A parent or guardian provides informed, written consent.
* A child 13 years or older (at enrollment/beginning of the school year) who provides assent.

Exclusion Criteria:

No exclusion criteria included in this protocol.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 5-16 year old children with complaints consistent with pharyngitis attending 4 public schools in Bamako, Mali.
Sampling Method: Non-Probability Sample
Enrollment: 1757 (Actual)
Dates: Start 2006-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The proportion of each emm-type among children with GAS pharyngitis. | Baseline day 0 through 3 year study period.

SECONDARY OUTCOMES:
Proportion of children with GAS pharyngitis who experience symptoms such as fever, exudative pharyngitis, tender cervical adenopathy, or scarletiniform rash, overall and by age in years. | Baseline day 0 through 3 year study period.
The incidence density (number of cases per children-weeks of follow up) of GAS pharyngitis among enrolled school children overall and according to: age in years, year of study, and season (cold or dry). | Baseline day 0 through 3 year study period.
The minimal incidence of GAS pharyngitis per 100,000 children in the catchment area of Djikoroni-para-Sébénikoro overall and according to: age in years, gender, year of study, and season (cold or dry). | Baseline day 0 through 3 year study period.
The proportion of each emm-type among children with GAS pharyngitis overall and according to: age in years, year of study, and season (cold or dry). | Baseline day 0 through 3 year study period.
The proportion of children with pharyngitis from whom GAS is isolated. | Baseline day 0 through 3 year study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Vaccine Development - Mali, Bamako, Bamako, Mali